CLINICAL TRIAL: NCT06146517
Title: A Single-Arm, Virtual Clinical Trial to Evaluate the Effects of a Sleep Supporting Beverage and Two Coffee Substitute Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clevr Blends (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20341
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Sleep; Mood; Caffeine Withdrawal; Anxiety; Productivity
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clevr Blends Arm (Experimental): Weeks 1-4: Participants will take one 6 oz serving daily of Clevr Blends Sleeptime 20 - 60 minutes before bed. The product comes with a scoop that measures 3 tsp. Participants should mix a full scoop with 6oz of water and froth using the frother that will be provided.
  Weeks 5-8: Participants will take one serving daily of Clevr Blends Matcha, before 1pm. The product comes with a scoop that measures 3 tsp. Participants should mix a full scoop with 6oz of water and froth using the frother that will be provided.
  Weeks 9-12: Participants will take one serving daily of Clevr Blends Chai, before 1pm. The product comes with a scoop that measures 3 tsp. Participants should mix a full scoop with 6oz of water and froth using the frother that will be provided.
  Interventions: Other: Clevr Sleeptime; Other: Clevr Matcha; Other: Clevr Chai

INTERVENTIONS:
Other: Clevr Sleeptime — Participants will trial Clevr Blends Sleeptime during weeks 1-4.
Other: Clevr Matcha — Participants will trial Clevr Matcha during weeks 5-8.
Other: Clevr Chai — Participants will trial Clevr Chai during weeks 9-12.

SUMMARY:
This is a virtual, single-arm clinical trial that will last 12 weeks. Participants will trial three different products, each for 4 weeks. Participants will trial Clevr Blends Sleeptime during weeks 1-4, Clevr Matcha for weeks 5-8, and Clevr Blends Chai for weeks 9-12. Participants will complete questionnaires at Baseline and Week 2, 4, 6, 8, 10, and 12. In addition to data will be collected from participants' sleep tracking devices at Baseline, Week 2, and Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Age 28-42.
* Generally healthy without any uncontrolled or chronic disease.
* Must consume a beverage containing low to moderate amount of caffeine once daily, defined as consuming the caffeine equivalent of less than or equal to one cup of coffee daily.
* Looking for healthier alternatives to caffeine.
* Currently owns a wearable sleep tracking device (e.g. Fitbit, Whoop, Oura etc) and has been wearing consistently for 4 weeks.
* Resident of the USA.

Exclusion Criteria:

* Allergies to any of the ingredients in the three products.
* Anyone with a formal diagnosis of insomnia.
* Any pre-existing or chronic conditions that would prevent participants from adhering to the protocol.
* Women that are pregnant, breastfeeding or attempting to conceive during the duration of the trial.
* Unwilling to follow the protocol.
* Participants that consume more than two caffeinated drinks daily.
* Participants that have little to no caffeine daily, equivalent to less than 1 cup of coffee daily.
* Is not a resident of the USA.

Ages: 28 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Change in sleep quantity as recorded by wearable sleep tracking device. [Timeframe Baseline to Week 4] | 4 weeks
  All participants will wear a sleep tracking device (e.g. Fitbit, Whoop, Oura etc) to record their total time asleep each night.
Changes in scores on the Sleep Quality Scale (SQS). [Timeframe Baseline to Week 4] | 4 weeks
  Consisting of 28 items, the SQS evaluates six domains of sleep quality: daytime symptoms, restoration after sleep, problems initiating and maintaining sleep, difficulty waking, and sleep satisfaction. Using a four-point, Likert-type scale, respondents indicate how frequently they exhibit certain sleep behaviors (0 = "few," 1 = "sometimes," 2 = "often," and 3 = "almost always").
Changes in self-reported energy levels. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires. Participants will answer on a Likert scale (0-5) with 0 indicating the best score and 5 indicating the worse score.
Changes in self-reported cognitive function. [Timeframe: Baseline to Week 12] | 12 weeks
  Measured via study-specific questionnaires. Participants will answer on a Likert scale (0-5) with 0 indicating the best score and 5 indicating the worse score.

SECONDARY OUTCOMES:
Changes in self-reported caffeine side effects, | 12 weeks
  Measured via study-specific questionnaires reviewing jitters, caffeine crashes, anxiety, negative moods and dependency. Participants will answer on a Likert scale (0-5) with 0 indicating the best score and 5 indicating the worse score.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided